CLINICAL TRIAL: NCT06364332
Title: Testing the Impact of #ChatsafeNL in a Randomized Controlled Trial: Does a Social Media Intervention Improve Dutch Young People's Safe Online Communication About Suicide?
Brief Title: Chatsafe Netherlands: Improving Safe Suicide Communication for Young People on Social Media
Acronym: CSNL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 113 Suicide Prevention (Other)
Collaborators: Orygen (Other); Mind (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ChatsafeNL; 2023.0348 (Other: Medical Ethics Committee VUmc)
Record Dates: First submitted 2024-04-02; First posted 2024-04-15 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Suicide Prevention; Communication; Social Media
Keywords: Suicide prevention; Suicidal Ideation; Communication; Social Media
MeSH Terms: conditions — Suicide Prevention; Communication; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Participants are randomized to the intervention or the control group using block randomization with varying block sizes (block sizes vary from 2 to 16). The distribution key will be 1:1. The randomization schedule is computer generated by a researcher who will not be part of the analysing researchers.
Who Masked: Investigator
Masking Description: The research team will be kept blind to randomization. A safety procedure is drawn up in which a senior researcher is appointed who will be unblinded if absolutely necessary. Principally, this will not be needed, since the study psychologists are independently alerted when a subject wants to get in touch.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): #Chatsafe suicide prevention content.
  Interventions: Behavioral: Social Media campaign
- Control (Active Comparator): Sexual health and wellbeing content
  Interventions: Behavioral: Social Media campaign

INTERVENTIONS:
Behavioral: Social Media campaign — Participants receive content three times a week; in total 24 pieces of content in 8 weeks. The content can consist of one or more photos or images with a caption (explanation in text).

SUMMARY:
Suicide is the leading cause of death among young people (YP) aged 10 to 25 years in the Netherlands. In addition, YP report high rates of suicidal ideation (16%). While suicidal behavior is a complex phenomenon with many factors and causes, the role of social media is becoming more prominent, especially for YP. Social media has been shown to be a source where YP can find support, but it's also a place where suicidal behavior is glorified or normalized, which can be triggering or harmful to other social media consumers.

The #Chatsafe guidelines were developed by Orygen Australia to better equip young people to communicate safely about suicide on social media. These guidelines are supported by a social media campaign to make the content of the guidelines more accessible to them. The #Chatsafe intervention consists of both the guidelines and the social media campaign. A small-scale Australian feasibility study showed promising results in terms of the acceptance and safety of the campaign, and safety regarding communicating about suicide on social media platforms. Currently, in Australia it is tested to what extent these results hold up in a Randomized Controlled Trial (RCT) (Robinson et al., 2023).

With funding from the Dutch National Agenda for Suicide Prevention, a contextualized replication study is conducted. The aim of this study is to determine whether the #Chatsafe intervention has an effect on the way in which Dutch YP communicate online about suicide.

DETAILED DESCRIPTION:
The #Chatsafe guidelines were developed by Orygen to better equip YP to communicate safely about suicide on social media. These guidelines are supported by a national social media campaign to make the content of the guidelines more accessible to the target group. The #Chatsafe intervention consists of both the guidelines and a social media campaign. A small-scale Australian feasibility study showed promising results in terms of acceptance and safety of the campaign, as well as the willingness of young people to intervene against suicide, their perceived self-efficacy, confidence, and safety regarding communicating about suicide on social media platforms. To test whether the effects hold up in a controlled setting, a Randomized Controlled Trial (RCT) is conducted.

With funding from the Dutch National Agenda for Suicide Prevention, commissioned by 113 Suicide Prevention, the #Chatsafe campaign is being translated to fit the Dutch context through a co-design process involving end users. To investigate whether this campaign has the intended effect in the Netherlands, a contextualized replication study into the efficacy of ChatsafeNL (Chatsafe Netherlands) is conducted in a controlled setting. The aim of the research is to determine whether the #ChatsafeNL intervention affects how YP, both with and without suicidal ideation, communicate online about suicide. A group receiving #ChatsafeNL content (intervention group) will be compared with a group who received content about sexual health and wellbeing (control group).

In the current study, the efficacy of the #ChatsafeNL intervention is tested in an RCT. The intervention condition (#ChatsafeNL social media intervention) is compared with a control intervention (sexual health campaign). The intervention phase lasts 8 weeks. Participants will be recruited over a period of 6-12 months.

Participants are asked to complete a self-report questionnaire at three different times, namely prior to the intervention (baseline, T1), immediately after the 8-week intervention (T2) and 4 weeks post-intervention (T3). During the intervention period, participants receive campaign content every week for 8 weeks. They are offered a short questionnaire to monitor safety and assess the evaluation of the content.

Initially, the campaign is developed for Instagram. This may expand to other social media platforms later on.

ELIGIBILITY:
Inclusion Criteria:

* age between 16-25 years,
* living in the Netherlands and speaking Dutch,
* see themselves as active social media user,
* is willing to share mobile phone number with the research team.

Exclusion Criteria:

None, if participants meet the inclusion criteria, they can principally participate in the study; having suicidal ideation is not a reason for exclusion. An extensive safety procedure is drawn up, which describes how the safety of the participants is monitored.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Safe communication about suicide online | Before, immediately after intervention and at 4 week follow up
  This outcome measure was specially developed for the Chatsafe Australia study, it will be measured by the purpose-designed #Chatsafe online safety questionnaire (Robinson et al., 2023) immediately after intervention. It is based upon an adapted version of the Perceived Safety Questionnaire.
  It consists of 4 different subscales, for each of which a sum score will be calculated: general use, seeing content, responding to content and interacting with content on social media. Overall sum score on communicating about self-harm and suicide on social media (25 items) ranges from 25-100, where higher scores reflect more safe communication.
  In addition, vignettes will be used to calculate scores concerning: sharing experiences of suicide online score, responding online to someone at risk and communication online about a suicide that has occurred (range 53-265). Here, also higher scores reflect more safe communication.

SECONDARY OUTCOMES:
Confidence when communicating about suicide online | Before, immediately after intervention and at 4 week follow up
  measured by the #Chatsafe online safety questionnaire
Willingness to intervene against suicide online | Before, immediately after intervention and at 4 week follow up
  measured via the Willingness to Intervene Questionnaire
Self-efficacy online | Before, immediately after intervention and at 4 week follow up
  measured by the Internet Self-Efficacy Questionnaire
Safety of the #ChatsafeNL materials | Before, immediately after intervention and at 4 week follow up
  measured by the weekly evaluation survey
Acceptability of the #ChatsafeNL intervention | Before, immediately after intervention and at 4 week follow up
  measured by the evaluation questions
Safety of the #ChatsafeNL intervention | Before, immediately after intervention and at 4 week follow up
  This is measured, among other things, by the number (or absence of) adverse events during the study period, such as a response to item 9 of the Patient Health Questionnaire that indicates they experience suicidal ideation, a response to the weekly questionnaire indicating that participants find the content disturbing, responses to the questionnaire that indicates that certain campaign content distressed participants and whether the research team was contacted by respondents to report distress or risk of self-harm or suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Mérelle, dr, Principal Investigator — 113 Suicide Prevention
Locations (1):
- 113 Suicide Prevention, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
The data will be made available upon reasonable request

REFERENCES:
- [Background] Robinson J, La Sala L, Cooper C, Spittal M, Rice S, Lamblin M, Brown E, Nolan H, Battersby-Coulter R, Rajaram G, Thorn P, Pirkis J, May-Finlay S, Silenzio V, Skehan J, Krysinska K, Bellairs-Walsh I. Testing the Impact of the #chatsafe Intervention on Young People's Ability to Communicate Safely About Suicide on Social Media: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Feb 17;12:e44300. doi: 10.2196/44300. PMID 36800220
- [Background] La Sala L, Pirkis J, Cooper C, Hill NTM, Lamblin M, Rajaram G, Rice S, Teh Z, Thorn P, Zahan R, Robinson J. Acceptability and Potential Impact of the #chatsafe Suicide Postvention Response Among Young People Who Have Been Exposed to Suicide: Pilot Study. JMIR Hum Factors. 2023 May 19;10:e44535. doi: 10.2196/44535. PMID 37204854
- [Background] La Sala L, Teh Z, Lamblin M, Rajaram G, Rice S, Hill NTM, Thorn P, Krysinska K, Robinson J. Can a social media intervention improve online communication about suicide? A feasibility study examining the acceptability and potential impact of the #chatsafe campaign. PLoS One. 2021 Jun 15;16(6):e0253278. doi: 10.1371/journal.pone.0253278. eCollection 2021. PMID 34129610